CLINICAL TRIAL: NCT04380506
Title: Drain Amylase Levels After Pancreatoduodenectomy. Validations of New cut-of for the Stratification of Postoperative Complications, Surgical Drains Management and Use of Postoperative Abdominal CT: (The DALCUT) Trial
Brief Title: Validations of New cut-of for the Stratification of Postoperative Complications,Drains Management
Acronym: DALCUT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Damiano Caputo, Associate Professor of Surgery, Campus Bio-Medico University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24/20 PAR ComEt CBM
Record Dates: First submitted 2020-04-21; First posted 2020-05-08 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Pancreas Cancer; Pancreatic Fistula
Keywords: Surgical Drain Managment; Pancreatic Fistula; Postoperative Complication; Amylase Drain level
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Fistula; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Drain removal (Experimental): Patients that fulfill criteria for surgical drains removal
  Interventions: Procedure: Surgical Drains Management

INTERVENTIONS:
Procedure: Surgical Drains Management — The Role of Amylase Drain Level in the Management of Surgical Drains after Pancreratoduodenectomy

SUMMARY:
Pancreatic fistula (PF) represents the Achille's heel of pancreatic surgery and is the main cause of postoperative morbidity since it can determine the onset of others complications such as abdominal abscesses, surgical wound infections, sepsis and bleeding, that can sometimes be fatal.

During a previous study conducted at the University Campus Bio-Medico of Rome, Department of General Surgery there were identified cut-offs of amylase levels on the abdominal drainage fluid dosed in I postoperative day (POD1) and III postoperative day (POD3) which can significantly predict PF and in particular clinically relevant fistulas as well as abdominal collections and biliary fistulas, if related to some specific findings of the abdominal CT routine performed in POD3.

The aim of this research project is to validate the cut-offs of the amylase levels on drainage fluid identified during the previous research in order to identify patients at risk of clinically relevant PF and to validate the use of abdomen CT without contrast in POD3 in patients with increased risk of biliary fistula.

DETAILED DESCRIPTION:
Pancreatic Fistula (PF) remains the main complication following pancreatic surgery with an incidence described in up to 45% of cases, even in high volume centers. It can determine the onset of other complications such as abdominal abscesses, surgical wound infections, sepsis and bleeding, sometimes fatal. In addition, the economic impact due to the extension of hospital stay and the management costs of the PF are not of secondary importance.

The International Study Group on Pancreatic Fistula (ISGFP) has standardized the definition of PF identifying it as "the leak from a surgical or percutaneous drainage of any measurable quantity of fluid, starting from the third postoperative day (POD3), with an amylase content three times higher than the upper normal limit of serum amylases. " However, according to this definition, all patients who satisfy this condition, even in the absence of any clinical signs or symptoms, are defined as suffering from pancreatic fistula.

To overcome this, a three grades classification system of PF was introduced, based on the clinical impact:

* Grade A: It is biochemical fistula; No intervention needed, not significant change of the post-operative hospital stay.
* Grade B: it requires an extension of the post-operative hospital stay, the permanence of surgical drains, the possible positioning of further drainages under radiological guide, antibiotic therapy and the use of artificial, enteral or parenteral nutrition;
* grade C: re-surgery is needed. Grade B and C represent clinically relevant fistulas. It is therefore evident that a correct definition of PF and its grade (A, B, C) can only be formulated "a posteriori".

However, considering the high prognostic impact of PF, it is needful to identify risk factors and diagnostic tools capable of stratifying patients at risk of pancreatic fistula and reach an early diagnosis in order to plan better plan both the treatment of it and the complications that may arise.

Many authors assume that the main predictive factor of PF is represented by the level of amylases in the abdominal drainage fluid, at different cut-offs and on different postoperative days. Others assume that abdominal drainage itself determines the development of PF and other complications.

Molinari has shown that a level of amylase in the abdominal drainage fluid <5000 IU / L in POD1 identifies a subgroup of patients at low risk of PF in which abdominal drainage is unfavorable to maintain. In Molinari's work, however, patients with PF grade A were also considered.

In his experience, Fong has identified a high-risk of PF subgroup in patients underwent DCP with an amylase level in abdominal drainage fluid > 600 IU / L in POD1. The author therefore proposed the immediate removal of abdominal drainage in patients considered low risk.

One of the most consistent bias of the Fong study is that in some patients there was an intrapancreatic drainage connected to the outside. Recently, Seykora has shown how in patients underwent DCP it is possible to use different amylase level cutoffs on drainage fluid in POD1, POD3 and POD5 in order to predict the clinically relevant PF risk and modulate the management of surgical drainages.

One of the limitations of the cut-offs identified by Seykora is represented by the fact that they have been identified considering their negative predictive value rather than their positive predictive value.

In a study recently conducted at Campus Bio-Medico University of Rome, Caputo confirmed that the dosage of amylase on the abdominal drainage fluid represents the most important clinically relevant predictor of PF and has confirmed, as underlined by Seykora, that the management of abdominal drainage is necessarily a dynamic process conditioned mainly by the serial dosage of amylases on drainage liquid (POD1-3).

Furthermore, in the Caputo's work, cut-offs of amylases on the abdominal drainage liquid (> 666 IU / L in POD1 and> 252 IU / L in POD3) have been identified as able to predict more than 80% of the clinically relevant PF. It has also been shown that the value of the amylases on the abdominal drainage fluid in POD3> 207 IU / L and the presence of an abdominal collection of dimensions equal to or greater than 5 cm in the abdomen CT without contrast performed on the same day significantly correlates with the risk of developing a biliary fistula.

If confirmed by this study, the practice of maintaining drainage in place up to POD3 could be validated. Drainages could be removed in POD3 in case of amylase levels in POD1 <666 U / L and amylase levels in POD3 <252 U / L except in cases where the amylase levels in POD3 are ≥ 207 and for which the routine use of abdominal CT on the same day seems to be justified in order to detect abdominal collections ≥ 5 cm which confirm the risk of this complication. In this latter category of patients, considering the risk of biliary fistula, drainages could be maintained beyond POD3.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old
* acquisition of informed consent for surgery and for inclusion in the study;
* elective open or laparoscopic PD

Exclusion Criteria:

* age <to 18 years;
* absence of informed consent for inclusion in the study;
* Emergency surgery;
* other pancreatic resections (not PD).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2020-03-15 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Validate the cut-offs of the amylase levels on drainage fluid identified during the previous research in order to identify patients at risk of clinically relevant FP | From postoperative day 1 to postoperative day 90
  The management of drainages and the execution of the abdomen CT scan in Postoperative day 3 will be managed on the basis of the outcome of the assay of amylase levels performed on fluid collected by surgical drains. This evaluation will be performed each day in the first three postoperative days or until drains removal.
Validate the ability of the diameter (in cm) of abdominal collection detected during the contrast-free abdomen CT in POD3 to predict risk of biliary fistula | From postoperative day 1 to postoperative day 90
  The relation between abdominal collections (measured in centimeters) detected with abdomen CT scan and the risk of develop a biliary fistula.

CONTACTS AND LOCATIONS:
Overall Officials: Damiano Caputo, MD, Principal Investigator — Campus Bio-Medico University
Locations (1):
- University Hospital Campus Bio-Medico of Rome, Roma, Italy

IPD SHARING:
Plan to Share IPD: No